CLINICAL TRIAL: NCT01492335
Title: Cognitive Assessment of Elderly Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PCP-AG023129
Record Dates: First submitted 2011-12-02; First posted 2011-12-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive decline; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Report (Experimental): Primary care physicians in the Cognitive Report group receive the results of their patients cognitive testing together with clinical diagnosis (Normal, Mild Cognitive Impairment, Dementia) and treatment recommendations.
  Interventions: Behavioral: Cognitive Report
- Treatment As Usual (Experimental): Physicians in the Treatment As Usual Group do not receive the results of their patients cognitive assessment, they do not receive treatment recommendations, nor are they told of the patients diagnosis (Normal, Mild Cognitive Impairment, Dementia)
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Cognitive Report — Physicians in the Cognitive Report group receive the results of their patients cognitive assessment which includes a clinical diagnosis (Normal, Mild Cognitive Impairment, Dementia) and treatment recommendations
  Arms: Cognitive Report
Behavioral: Treatment As Usual — Physicians in the Treatment As Usual group do not receive the results of their patients cognitive assessments, they are not given treatment recommendations nor are they told of the patients clinical diagnosis (Normal, Mild Cognitive Impairment, Dementia).
  Arms: Treatment As Usual

SUMMARY:
Most primary care physicians do not screen older patients for cognitive impairment. Identification of cognitive impairment may result in earlier referral for diagnostic work-up and earlier treatment and better patient outcomes. The purpose of this study is to determine whether physicians who receive the results of a cognitive screen use this information in treatment plans and whether this results in better cognitive outcomes for the older patients.

DETAILED DESCRIPTION:
Current trends in healthcare suggest that in the coming decade most older patients will obtain services solely through the general practice/family practice sector of healthcare. Effective and optimal management of older patients with multiple complex medical conditions and compromised cognitive functioning will be a challenge for the primary care physician (PCP). Early identification of older patients with cognitive deficits should allow early referral for diagnostic work-up and earlier treatment and better patient outcomes. The goal of this study is to investigate the utility of providing cognitive testing in the PCP office. PCPs will be randomized to either Treatment As Usual (TAU) or Cognitive Report (CR). The study hypotheses are (1) patients of physicians in the CR group will have improved clinical outcomes i.e. cognitively impaired patients in the CR group will have a slower rate of progression of cognitive deficits over two years than cognitively impaired patients in the TAU group; (2) PCPs in the CR group will order dementia screening tests, refer to specialists and prescribe anticholinesterase inhibitors more frequently than PCPs in the TAU group.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over
* Plan to remain a patient of this physician for two years
* MMSE score greater than 18

Exclusion Criteria:

* Diagnosis of Dementia, Alzheimer's disease, Huntington's disease, Vascular disease or other dementing disorder
* MMSE score of 18 or less
* Sensory deficit e.g. limited vision or hearing precluding cognitive testing

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 524 (Actual)
Dates: Start 2006-01; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Scores on a comprehensive battery of neuropsychological tests. | Two years
  Diagnosis is based on performance on a standard neuropsychological test battery that assesses mutliple cognitive domains known to be sensitive to early dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Saxton, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States